CLINICAL TRIAL: NCT05041478
Title: Cold Snare Endoscopic Mucosal Resection vs Cold Snare Endoscopic Mucosal Resection With Adjuvant Thermal Therapy to Resection Margins - A Randomised Controlled Trial
Brief Title: Cold Snare Endoscopic Mucosal Resection (EMR) vs Cold EMR With Margin Snare Tip Soft Coagulation (STSC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Professor, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETH11029
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Polyp; Colon Adenoma; Colon Cancer
Keywords: Colonoscopy; Polypectomy; Adenoma; Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Adenoma; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold EMR with adjuvant STSC to margins (Experimental): Standard cold EMR technique with adjuvant snare tip soft coagulation to defect margins
  Interventions: Procedure: Cold Snare Endoscopic mucosal resection with adjuvant snare tip soft coagulation
- Cold EMR (Active Comparator): Standard Cold EMR resection technique
  Interventions: Procedure: Cold Snare Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Cold Snare Endoscopic mucosal resection with adjuvant snare tip soft coagulation — Use of injected chromogelofusine solution to raise a lesion prior to polypectomy. Lesion then removed with a stiff thin-wired snare. Following this defect margins are treated with electrocautery to create a rim of ablated tissue.
  Arms: Cold EMR with adjuvant STSC to margins
Procedure: Cold Snare Endoscopic Mucosal Resection — Use of injected chromogelofusine solution to raise a lesion prior to polypectomy. Lesion then removed with a stiff thin-wired snare.
  Arms: Cold EMR

SUMMARY:
Randomised controlled trial comparing cold snare endoscopic mucosal resection (EMR) with cold snare EMR and adjuvant margin STSC in the complete resection of 15-40mm lateral-spreading adenomas

DETAILED DESCRIPTION:
Rationale:

Conventional EMR is well-established for the resection of lateral-spreading adenomas and has been shown to be highly efficacious with adjuvant STSC. Cauterisation-related complications occur relatively frequently and while endoscopically treatable, still carry morbidity not seen in current cold snare polypectomy data.

Cold snare polypectomy has an excellent safety profile for smaller polyps, without cauterisation-related adverse events. Limited data on cold EMR for large adenomatous laterally-spreading lesions shows minimal complications. Efficacy, however, is yet to be evaluated in prospective randomised trials. Observational data demonstrates recurrence rates exceeding conventional EMR. Since STSC causes significant reduction in recurrence in conventional EMR, the safety and efficacy of this adjuvant technique, when compared to isolated cold snare EMR, has theoretical advantages in both safety and efficacy.

The safety and efficacy of these two techniques will therefore be compared in a randomised controlled trial.

Hypothesis:

Cold snare EMR of 15-40mm lateral-spreading adenomas with adjuvant STSC is expected to be superior regarding complete resection and adenoma recurrence rates as compared to cold snare EMR.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing colonoscopy who is older than 18 years of age, has a written consent for trial participation and has at least one laterally spreading lesion meeting the following description:
* Localisation in the colon or rectum
* Benign adenomatous surface features (Kudo III / IV, Japan NBI Expert Team (JNET) 2a)
* Granular or non-granular topography
* Paris classification 0-IIa/IIb +/- Is
* If present, sessile component may be no greater than 10mm in size.
* Polyp size ranging from 15 to 40mm

Exclusion Criteria:

* Current use of antiplatelet (excluding aspirin) or anticoagulants which have not appropriately been interrupted according to the guidelines.
* Known bleeding disorder or coagulopathy.
* Pregnancy
* History of inflammatory bowel disease
* Previously attempted or otherwise non-lifting lesions
* Endoscopic features suggestive of submucosal invasion (Kudo Vi/n, JNET 2b / 3) or concurrent colorectal cancer
* Lesions involving the ileocaecal valve (ICV), appendiceal oriface or anorectal junction (ARJ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete resection rate (CRR) | 1 day
  Determined by endoscopic assessment (no visible residual adenoma) and histological assessment (biopsies of resection margin)
Adenoma recurrence rate (ARR) | 4-6 months
  ARR at first surveillance colonoscopy (SC1) as determined by endoscopic assessment (no visible recurrent adenoma) and histological assessment (scar biopsies)

SECONDARY OUTCOMES:
Intra-procedural and post-procedural complication rates | 30 days
  Intraprocedural bleeding, clinically significant post-polypectomy bleeding, deep mural injury, post polypectomy coagulation syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, Principal Investigator — Westmead Hospital (WSLHD)
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia